CLINICAL TRIAL: NCT05581654
Title: Vaginal Natural Orifice Trans-luminal Endoscopic Surgery (vNOTES) Salpingectomy for Tubal Sterilization: Clinical Outcomes and Learning Curve Analysis: A Multicentre Prospective Study
Brief Title: Vaginal Natural Orifice Trans-luminal Endoscopic Surgery Salpingectomy for Tubal Sterilization: Clinical Outcomes and Learning Curve Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jani Jacques (Other)
Responsible Party: Sponsor-Investigator, Jani Jacques, Head of Gyneco-Obstetrics Department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LC-V-NOTES
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Tubal Sterilization
MeSH Terms: interventions — Salpingectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Junior surgeons (Experimental): The surgeons will be divided into 2 arms based on their surgical experience time: less than 5 years (junior surgeons) and more than 5 years (senior surgeons). The learning curve analysis will include 30 procedures for each surgeon group in each centre. For ethical reasons, all the junior surgeons will first assist the senior surgeons in performing vNOTES salpingectomy, as first assistant in at least 15 procedures, before starting to perform them as operators.
  Interventions: Procedure: Salpingectomy
- Senior surgeons (Active Comparator): The surgeons will be divided into 2 arms based on their surgical experience time: less than 5 years (junior surgeons) and more than 5 years (senior surgeons). The learning curve analysis will include 30 procedures for each surgeon group in each centre.
  Interventions: Procedure: Salpingectomy

INTERVENTIONS:
Procedure: Salpingectomy — Salpingectomy by vaginal natural orifice transluminal endoscopic surgery (v-NOTES).

SUMMARY:
The evolution from classical open surgery to laparoscopic surgery has led to a significant reduction of morbidity and mortality.

Newer advances such as development of single port laparoscopic surgery and scarless Natural Orifice Transluminal Endoscopic Surgery (NOTES) have moved forward the practice in "Minimally Invasive Surgery".

Recently, clinical application of vNOTES has broadened significantly in the field of gynaecological surgery.

As the application of vNOTES is increasing, it is deemed mandatory to assess the clinical outcomes and the learning curve (LC) of this novel technique.

There is a paucity of reports in the literature analysing prospectively the clinical outcomes the LC of vNOTES in the gynaecological field.

To the investigator's knowledge, there is no published prospective multicentre study that aims to evaluate the peri- and postoperative outcomes and the LC of salpingectomy for tubal sterilization by the technique of vNOTES.

DETAILED DESCRIPTION:
The evolution from traditional open surgery to laparoscopic surgery has led to a significant reduction of morbidity and mortality. Newer advances such as development of single port laparoscopic surgery and scarless Natural Orifice Transluminal Endoscopic Surgery (NOTES) with or without robot assistance have moved forward the practice in "Minimally Invasive Surgery".

Described for the first time in 2004 at John Hopkins University in an experimental porcine model, NOTES is a surgical technique in which the natural orifices (mouth, vagina, urethra and rectum) are used as access routes to the peritoneal cavity for endoscopic surgery with no abdominal incisions.

Clinical application of NOTES has been initially reported in general surgical procedures where Trans-gastric Appendectomy and Cholecystectomy have been performed using the mouth and the stomach as the access route.

The technique seems to be feasible and safe when performed by experienced surgeons. Favourable outcomes such as reduced post-operative pain, a shorter length of hospital stay, improved cosmetic results due to scar-free surgery and reduced wound complications at trocar insertion sites, promote the increasing use of this new surgical technique.

Although NOTES may be performed through various entries including the stomach, oesophagus, bladder and rectum, NOTES procedures in women have been commonly performed through the vagina as this allows direct access to the abdominal cavity. Therefore, trans-vaginal NOTES (vNOTES) has gained popularity among general surgeons, urologists and gastroenterologists over the past decade and was adopted in various surgical procedures, varying from cholecystectomy, appendectomy, sigmoidectomy, nephrectomy, splenectomy, liver resection and sleeve gastrectomy.

Recently, clinical application of vNOTES has broadened significantly in the field of gynaecological surgery. The feasibility and safety of vNOTES in this specialty was firstly demonstrated in 2012. This event represented the key milestone in the evolution of vNOTES for gynaecologic procedures. Based on the current reports, we know that many of these procedures, such as oophorectomy, salpingectomy, adnexectomy, hysterectomy and many other more complex surgeries can be performed using vNOTES by the majority of surgeons who have adequate skills in performing laparoscopy.

As the application of vNOTES is increasing, it is deemed mandatory to assess the learning curve (LC) of this novel technique. This is particularly important in surgery where new skills must be acquired constantly, safely and proficiently. It would be useful to know how many vNOTES procedures a surgeon may have to carry out before reaching an adequate level of safety and efficiency. Furthermore, a correct understanding of the LC is essential in randomised control trials comparing vNOTES with alternative types of surgery in order to reach valid conclusions.

There is a paucity of reports in the literature analysing the LC of vNOTES. The "learning curves" for performing vNOTES hysterectomy and adnexal surgery have been previously assessed by retrospective studies, each conducted on a single surgeon basis and in a single institution (19-21). In a report published in June 2020, Lowenstein et al were among the first researchers that evaluated prospectively the learning curve of mastering the skills to perform vNOTES hysterectomy and uterosacral ligament suspension in two different centres.

To the investigators knowledge, there is no published prospective multicentre study that aims to evaluate the feasibility, the LC, the peri- and postoperative outcomes of salpingectomy for tubal sterilization by the technique of vNOTES.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 50 years
* Non-prolapsed uterus
* Asking for tubal sterilisation
* Any parity
* Written informed consent

Exclusion Criteria:

* History of pelvic inflammatory disease.
* Recto-vaginal endometriosis.
* Suspicion of genital tract malignancy.
* Active lower genital tract infection.
* History of rectal surgery.
* Stage III or IV Uterine prolapse (defined by the International Continence Society classification).
* Complete obliteration of the posterior douglas pouch determined by pelvic examination.
* Virginity.
* Failure to provide written informed consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of women successfully operated (salpingectomy) for tubal sterilization using vNOTES technique as a one day procedure. | 2 years
  The proportion of women who were successfully operated (salpingectomy) for tubal sterilization using vNOTES technique as a one day procedure will be measured as the primary outcome of effectiveness.
  Successful salpingectomy for tubal sterilization using vNOTES technique as a one day procedure is defined by:
  * Complete retrieval of fallopian tube(s) (pathological confirmation).
  * No conversion into laparoscopy or open surgery.
  * Discharge from hospital on day 0 post-operatively.
Learning Curve Assessment. | 2 years
  The Assessment of the learning curve of salpingectomy by the technique of vNOTES in young and experienced surgeons is another primary outcome of our study.

SECONDARY OUTCOMES:
Intraoperative or postoperative complications | 6 weeks
  Intraoperative or postoperative complications detected during the first 6 weeks of surgery and classified based on the Clavien-Dindo classification.
Postoperative pain scores | 7 days
  Postoperative pain scores measured using a visual analog scale twice a day from day 1 to 7.
Pain drugs intake | 7 days
  The total amount of pain drugs taken during the first week following surgery
Number of days of absence from work | 2 years
  Number of days of absence from work
Short Sexual Functioning Scale (SSFS) | baseline
  Sexual well-being by self-reporting the Short Sexual Functioning Scale (SSFS).
Short Sexual Functioning Scale (SSFS) | 3 months after baseline
  Sexual well-being by self-reporting the Short Sexual Functioning Scale (SSFS).
Short Sexual Functioning Scale (SSFS) | 6 months after baseline
  Sexual well-being by self-reporting the Short Sexual Functioning Scale (SSFS).
Pain on sexual intercourse | baseline
  Occurrence and severity of pain on sexual intercourse self-reported by the patient by using a simple questionnaire.
Pain on sexual intercourse | 3 months after baseline
  Occurrence and severity of pain on sexual intercourse self-reported by the patient by using a simple questionnaire.
Pain on sexual intercourse | 6 months after baseline
  Occurrence and severity of pain on sexual intercourse self-reported by the patient by using a simple questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros KARAMPELAS, MD, Principal Investigator — CHU Brugmann
Locations (4):
- Belgium (4):
  - Clinique Saint-Jean, Brussels
  - CHU Brugmann, Brussels
  - Cliniques Universitaires Saint LUC, Brussels
  - CHU Liège - site CHR Liège, Liège

IPD SHARING:
Plan to Share IPD: No